CLINICAL TRIAL: NCT00775723
Title: Term-Born Infants at 9 and 12 Months of Age: A Randomized Controlled Trial
Brief Title: Melatonin Production Delay in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Tel Aviv University (Other)
Responsible Party: Dr Sari Goldstein Ferber, Director of Developmental Care, Sackler School of Medicine Tel Aviv University
Other Study IDs: 1673; 0
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Melatonin Production
Keywords: 6sulphatoxymelatonin; preterm infants; melatonin is low in preterm infants at least until the age of 6 months

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: Melatonin production is known to be delayed in preterm-born infants up to 6 months of age. This might be related to exposure of preterm infants to continuous lighting in the NICU during a critical period of pineal gland development. The investigators aimed to test the profile of melatonin production in these infants at 9-12 months of age.

Methods: Twenty three term-born and 23 preterm-born infants (gestational age: 29-34 weeks) were studied. The investigators tested nocturnal urinary melatonin excretion, within a repeated measures design, both at 9 and 12 months of age. Nocturnal urine was extracted from diapers and urinary melatonin derivate (6-sulphatoxymelatonin) excretion was analyzed by ELISA assay.

DETAILED DESCRIPTION:
Unlike other organs which show catch up in preterm infants after one year of life, the pineal gland shows persistent delay in melatonin production. This field of research has been neglected lately although there are published recommendations for decrease of bright light in NICUs which prevents melatonin development and production, and also recommendations for melatonin treatment in cases respiration recovery in hospitalized preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* The investigators included healthy mothers with singleton pregnancies and documented prenatal care who were admitted before term (28-34) weeks gestation to the hospital's delivery room with early uterine contractions and entering stage 1 of an anticipated spontaneous vaginal delivery or term infants born at 38-42 weeks of gestation.

Exclusion criteria:

* Mothers who showed signs of fetal distress during labor, or required Cesarean (C)c-section, or had fetuses withand estimated fetal weights < 10th percentile for gestational age and children diagnosed with

  * Genetic anomalies, congenital heart malformations, gastrointestinal disturbances and central nervous system dysfunction
  * Age < 9 months, Age > 9 months month at onset of study
  * Considered medically unstable

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Design: Forty-six infants (23 full term and 23 preterm babies) infants and their mothers were randomly recruited from a successive list of preterm and term labors at a large urban medical center in Northern Israel and were assigned to the study. We calculated that a sample size of 30 mother-infant dyads is sufficient to show a significant effect of the intervention with a power of 90% and 5% risk of type alpha error (Cohen , chen, West & Aiken, 2003). This calculation was based on the effect size found in full-term infants melatonin secetion (1).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sari Goldstein Ferber, Study Director — Sackler School of Medicine, Tel Aviv Universitry
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Ferber SG, Laudon M, Kuint J, Weller A, Zisapel N. Massage therapy by mothers enhances the adjustment of circadian rhythms to the nocturnal period in full-term infants. J Dev Behav Pediatr. 2002 Dec;23(6):410-5. doi: 10.1097/00004703-200212000-00003. PMID 12476070
- [Background] Ferber SG, Makhoul IR. Neurobehavioural assessment of skin-to-skin effects on reaction to pain in preterm infants: a randomized, controlled within-subject trial. Acta Paediatr. 2008 Feb;97(2):171-6. doi: 10.1111/j.1651-2227.2007.00607.x. Epub 2008 Jan 3. PMID 18177441
- [Background] Ferber SG, Makhoul IR. The effect of skin-to-skin contact (kangaroo care) shortly after birth on the neurobehavioral responses of the term newborn: a randomized, controlled trial. Pediatrics. 2004 Apr;113(4):858-65. doi: 10.1542/peds.113.4.858. PMID 15060238